CLINICAL TRIAL: NCT01810471
Title: External Ankle Supports - 3D Motion Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Benita Kuni, MD, Principal Investigator, Job Title: Orthopedic and Trauma Surgeon, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 407- 05_130307
Record Dates: First submitted 2013-03-10; First posted 2013-03-13 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ankle supports (Experimental)
  Interventions: Device: Applying ankle support device (white non-elastic tape, kinesiotape (TM), soft brace (Malleotrain TM)

INTERVENTIONS:
Device: Applying ankle support device (white non-elastic tape, kinesiotape (TM), soft brace (Malleotrain TM)

SUMMARY:
Untreated ankle sprains often remain symptomatic and may end in chronic instability. The aim of our study is to quantify the stabilizing effect of different devices. Through the use of a foot measurement model in 3D motion analysis the influence of the devices with respect to a mechanical effect is examined by means of different tests. The dynamic postural control is quantified. The hypothesis was that the devices would stabilize differently the foot segments.

ELIGIBILITY:
Inclusion Criteria:

* chronic ankle instability
* "giving way"
* repeated ankle sprains

Exclusion Criteria:

* other injuries of the lower extremities
* surgery on the lower extremities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
change of the range of motion of the subtalar inversion/eversion in degree | baseline (=before) and immediately after applying the device

CONTACTS AND LOCATIONS:
Overall Officials: Benita Kuni, Dr. med., M.D., Principal Investigator — Dep. of Orthopedics, Trauma Surgery and Spinal Cord Injury
Locations (1):
- Department of Orthopedics, Trauma Surgery and Spinal Cord Injury, Heidelberg University Hospital, Heidelberg, Germany

REFERENCES:
- [Derived] Kuni B, Mussler J, Kalkum E, Schmitt H, Wolf SI. Effect of kinesiotaping, non-elastic taping and bracing on segmental foot kinematics during drop landing in healthy subjects and subjects with chronic ankle instability. Physiotherapy. 2016 Sep;102(3):287-93. doi: 10.1016/j.physio.2015.07.004. Epub 2015 Sep 3. PMID 26422550